CLINICAL TRIAL: NCT05887622
Title: The Role of Potassium Supplementation on Endothelial Function, BP Regulation, and Oxidative Stress Under High Sodium Conditions
Brief Title: The Potassium Supplementation Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Delaware (Other)
Responsible Party: Principal Investigator, Shannon Lennon, Associate Professor, University of Delaware
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: 1465208
Record Dates: First submitted 2022-03-29; First posted 2023-06-05 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2025-06

CONDITIONS: Cardiovascular Health; Cardiovascular Risk Factor

STUDY DESIGN:
Intervention Model Description: All participants will complete all arms in a randomized, crossover design.
Who Masked: Participant
Masking Description: Participants will be blinded to the diet they are on.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Moderate potassium/low sodium (Experimental): Subjects will consume a diet moderation in potassium and low in sodium.
  Interventions: Dietary Supplement: Placebo
- Moderate potassium/high sodium (Experimental): Subjects will consume a diet moderation in potassium and high in sodium.
  Interventions: Dietary Supplement: Placebo
- High potassium/high sodium (Experimental): Subjects will consume a diet moderation in potassium and high in sodium.
  Interventions: Dietary Supplement: Potassium chloride supplement

INTERVENTIONS:
Dietary Supplement: Potassium chloride supplement — Subjects will receive 64 mmol of KCl on the high potassium/high sodium condition.
  Arms: High potassium/high sodium
Dietary Supplement: Placebo — Subjects will receive a placebo capsule on the moderate potassium/low sodium diet and the moderate potassium/high sodium diet
  Arms: Moderate potassium/high sodium; Moderate potassium/low sodium

SUMMARY:
This study will test whether potassium supplementation can reduce the deleterious effect of a high sodium diet on blood vessel function, blood pressure reactivity and autonomic nervous system function in apparently healthy adults.

DETAILED DESCRIPTION:
Excess sodium intake is linked to poor blood pressure (BP) regulation and endothelial dysfunction, both of which are implicated in the pathogenesis of atherosclerosis and high BP. Evidence suggests potassium may offset the damaging effects of sodium; however, studies in healthy adults are lacking. This is important as these pre-clinical risk factors have been observed in this population, suggesting early intervention may be critical for cardiovascular disease prevention. High potassium diets have been effective at attenuating a sodium-induced decline in endothelial function. However, potassium intake was increased using whole foods; thus, the vascular benefits cannot be attributed solely to potassium. Furthermore, whether potassium can reduce sodium-induced oxidative stress is unknown. The central hypothesis of this study is that endothelial function will be greater and BP reactivity and oxidative stress will be lower with a high potassium intake compared to a low potassium intake, in the context of a high sodium diet. The investigators will assess macrovascular function using flow-mediated dilation, BP reactivity using the cold pressor test and isometric handgrip grip test, and oxidative stress using electron paramagnetic resonance.

ELIGIBILITY:
Inclusion Criteria:

* men and women
* 18-45 years of age
* all races/ethnicities
* BMI < 30 kg/m2
* BP < 130/80 mmHg

Exclusion Criteria:

* presence of hypertension
* known heart disease
* diabetes
* kidney disease
* cancer
* inflammatory conditions
* blood clotting disorders
* pregnancy
* adrenal gland disorder
* history of stomach or intestinal bleeding
* history of kidney stones
* serum potassium outside of the normal range

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-01-24 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
Conduit artery endothelial dependent dilation | on day 10 of each diet
  The difference in flow-mediated dilation (FMD) between the 3 diets
Blood pressure reactivity | on day 10 of each diet
  The change in both systolic and diastolic blood pressure during handgrip exercise and cold pressor test from baseline
Superoxide levels | on day 10 of each diet
  The difference in superoxide levels as measured by electronic paramagnetic resonance (EPR) between the 3 diets will be assessed

CONTACTS AND LOCATIONS:
Locations (1):
- Tower at STAR, Newark, Delaware, United States